CLINICAL TRIAL: NCT00832715
Title: Diagnostic Utility of Endobronchial Ultrasound Guided Mediastinal Lymph Node Sampling in Clinical Stage I and II Non Small Cell Lung Cancer
Brief Title: Utility of Endobronchial Ultrasound Guided Needle Biopsy in Early Stage Non- Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0387; NCI-2015-01900 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: Lung; Lung Cancer; NSCLC; Non Small Cell Lung Cancer; Squamous Cell; Adenocarcinoma; Large Cell; Endobronchial Ultrasound Transbronchial Needle Aspiration; Mediastinal lymph node negative disease; Mediastinal Nodal Metastasis; EBUS-FNA; Endobronchial Ultrasound Fine Needle Aspiration; EBUS guided needle mediastinal lymph node biopsy; Biopsy; PET scan; Positron Emission Tomography; CT Scans; Computed Tomography Scans; Lymph node; Mediastinoscopy; Bronchoscope
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBUS-TBNA (Experimental): Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA)
  Interventions: Procedure: EBUS-TBNA

INTERVENTIONS:
Procedure: EBUS-TBNA — Tissue sample collected bronchoscope using needle aspirate of lung lymph gland, procedure takes 1 hour.
  Other Names: Endobronchial Ultrasound Transbronchial Needle Aspiration

SUMMARY:
The goal of this clinical research study is to learn how accurately an endobronchial ultrasound transbronchial needle aspiration (EBUS -TBNA) may detect mediastinal lymph node metastases in patients with clinical stage I and II non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Study Procedures:

A procedure called EBUS-TBNA has been developed that might allow doctors to get samples of lymph glands without performing an operation. The standard practice is a surgical operation called a mediastinoscopy. If researchers find out that EBUS-TBNA is as accurate as mediastinoscopy, it may mean that patients with lung cancer can avoid having surgery or will be able to get treatment before surgery.

EBUS-TBNA:

If you agree to take part in this study, you will first have an EBUS-TBNA. This will be performed on an out-patient basis under general anesthetic. The doctor will examine your lungs for suspicious lymph glands with an ultrasound, and then will take a sample of tissue from the lymph gland. This will be done using a flexible scope called a bronchoscope that can be passed into the windpipe. The lymph glands around the wind pipe can be seen and then removed with a small needle. The procedure should take about 1 hour.

Researchers will then analyze the lymph glands that were removed. Depending on whether or not the lymph glands have cancer in them, your doctor will then recommend the most appropriate therapy for you. This may include mediastinoscopy or some other appropriate therapy.

All the data for the study will be stored with a password protected system.

Length of Study:

Your participation in this study will be over after you have completed EBUS-TBNA.

This is an investigational study. EBUS-TBNA is FDA approved for this procedure.

Up to 120 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be >/= 18 years old.
2. Patient must have Eastern Cooperative Oncology Group (ECOG)/Zubrod status 0-2.
3. Patient must have proven or suspected NSCLC (squamous cell, adenocarcinoma, or large cell) and be clinical Stage I or II, according to the 1998 staging system of the American Joint Commission on Cancer for lung cancer (T1-3 N0, T1-2 N1).
4. Patient must be eligible for definitive surgical therapy for primary NSCLC.
5. Patient or the patient's legally acceptable representative must provide written informed consent prior to registration and any study-related procedures.
6. If the patient is a survivor of a prior invasive cancer, all of the following criteria must apply: a. Patient has undergone potentially curative therapy for all prior malignancies. b. No evidence of active / recurrent disease.
7. All females of childbearing age must have a negative pregnancy test before beginning the study.

Exclusion Criteria:

1. Patient has received prior chemotherapy or radiotherapy for this cancer.
2. Patient is considered a poor risk for surgery due to non-malignant systemic disease (cardiovascular, renal, etc.) that would preclude the treatment options.
3. Patient has contraindication to either endobronchial ultrasound or mediastinoscopy such as: history of bleeding diathesis, latex allergy, mediastinoscopy, mediastinal nodal resection, tracheostomy.
4. Patients malignancy consistent with well differentiated (carcinoid) neuroendocrine histology.
5. Patient has two separate same histology lung tumors (where the question of two separate primaries or metastatic disease makes definitive clinical staging inaccurate).
6. Females who are pregnant and/or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with False Negative Rate Using EBUS Guided Mediastinal Lymph Node Biopsy | Patient participation 1 hour to complete EBUS-TBNA
  False negative rate estimated using EBUS guided mediastinal lymph node biopsy following a negative positron emission tomography (PET) scan with a 90% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: George A. Eapen, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org